CLINICAL TRIAL: NCT01414777
Title: IRB-HSR# 14583: Intravenous Ondansetron to Attenuate the Hypotensive, Bradycardic Response to Spinal Anesthesia in Healthy Parturients
Brief Title: Intravenous Ondansetron to Attenuate the Hypotensive, Bradycardic Response to Spinal Anesthesia in Healthy Parturients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Mohamed Tiouririne, MD, Associate Professor of Anesthesiology, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 14583
Record Dates: First submitted 2010-09-16; First posted 2011-08-11 (Estimated); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Hypotension; Pregnancy
Keywords: c-section; Hypotension after spinal anesthesia for C-section
MeSH Terms: conditions — Hypotension | interventions — Ondansetron; Injections, Epidural

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ondansetron (Experimental): ondansetron 8 mg IV will be administered prior to placement of the spinal anesthesia
  Interventions: Drug: ondansetron
- Placebo (Placebo Comparator): Ondansetron 8 mg IV or Placebo will be administered prior to placement of the spinal anesthestic
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ondansetron — Ondansetron 8mg IV or placebo will be administered prior to placement of the spinal anesthetic
  Other Names: epidural
  Arms: ondansetron
Drug: placebo — placebo or ondansetron 8mg IV will be administered prior to placement of the spinal anesthetic
  Other Names: epidural
  Arms: Placebo

SUMMARY:
The investigators hypothesize that given prophylactically, intravenous ondansetron will attenuate the drop in blood pressure and heart rate frequently seen after spinal anesthesia.

Eighty-six American Society of Anesthesiologists (ASA) physical status I or II in preoperative patient assessment, parturients age of 18 to 45 years scheduled to undergo elective caesarean section will be enrolled.

Patients will be randomized to 2 groups: the ondansetron group, receiving 8 mg intravenous ondansetron diluted in 10 mL of saline; or the placebo group, who were administered 10 mL of saline given 5 minutes prior to performing the spinal anesthetic. Investigational Pharmacy will randomize and dispense study drug.

Baseline measurements of vital signs will be taken. Otherwise standard management will then be used:

* Patients must be NPO for 8 hours
* Pulse oximetry, EKG monitoring, noninvasive blood pressure at a minimum of every 3 minutes, more frequently if decided by the provider.
* Standard lumbar puncture in a sitting position the L3-L4 or L4-L5
* Whitacre pencil-point, 25 gauge
* Injectate: 2 mL of 0.75% hyperbaric bupivacaine, 100 mcg preservative free morphine, 20 mcg fentanyl
* Immediately after completing the subarachnoid injection, patients will be laid supine with left lateral uterine displacement

The sensory level of anesthesia will be assessed in the standard fashion every five minutes using ice. The motor component will tested using the Bromage scale for spinal anesthesia (0, no paralysis; 1, inability to lift the thigh [only knee/feet]; 2, inability to flex the knee [only feet]; 3, inability to move any joint in the legs).

DETAILED DESCRIPTION:
Over the last 30 years, regional anesthesia has emerged as the method of choice for elective caesarean section because it avoids risks involved in managing the airway of the parturient and has the added significant benefit of mother being awake for the birth of her child. Indeed, this changing practice patterns is thought to have lead to a significant drop in anesthesia related maternal morbidity and mortality.

At the same time, regional anesthesia is associated with both minor and significant risk.

Most common among these effects is hypotension and bradycardia, occurring in 33% and 13% of cases, respectively. In the pregnant patient, supine positioning required for surgery is associated hypotension due to aortocaval compression by the gravid uterus in 8% of patients, even without spinal anesthesia. During caesarean section, the combination of these factors can lead to hypotension include decreased placental blood flow, impaired fetal oxygenation and fetal acidosis. Maternal symptoms of low blood pressures include nausea, vomiting, dizziness, and decreased consciousness. This situation has lead to dozens of publications seeking to prevent or minimize the hypotensive response.

Hypotension after a spinal is initially due to a blockade of sympathetic fibers leading to a drop in systemic vascular resistance. Spinal-induced bradycardia is multifactorial but is in part due to the Bezold-Jarisch Reflex (BJR). This reflex is mediated by serotonin receptors within the wall of the ventricle in response to systemic hypotension. These receptors, the 5HT3 subtype, cause an increase efferent vagal signaling when bound by serotonin released during hypovolemic states, clinically leading to bradycardia and further hypotension.

Ondansetron, a widely used anti-emetic and serotonin antagonist, has been safely used to blunt the BJR, resulting in less bradycardia and hypotension first in animals and later in humans undergoing spinal anesthesia. ,

Use During Pregnancy:

The FDA labels ondansetron as a class B. Studies in pregnant rats and rabbits at doses up to 70 times higher than clinically used doses revealed no evidence of impaired fertility or harm to the fetus due to ondansetron. There are, however, few prospective studies in pregnant women. Nevertheless, the drug is widely used has a long safety history for use in pregnancy and during anesthesia for caesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Elective Caesarean section
* Consent to be in the study
* Age 18-45
* ASA 1 or 2

Exclusion Criteria:

* Patient refusal
* Patients with known allergy to ondansetron will be excluded
* Contraindications to spinal anesthetic

  * Known Coagulopathy (acquired e.g. anticoagulation or existing such as liver disease; using patient history, physical examination to determine bleeding risks, a platelet count under 100 or a PT INR over 1.4)
  * Severely altered anatomy (e.g. post surgical changes)
  * Existing neurological deficits (Women with a history of migraine or tension headache will be allowed to enroll. More severe conditions with daily life limiting symptoms will be excluded. Examples include epilepsy, pseudotumor cerebri, prior stroke with persistent neurologic deficits, or any motor or sensory neuropathy with existing deficits)
  * Skin infection overlying site

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2009-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability" | day 1
  hypotension & bradycardia will be recorded from the placement of the spinal through the end of surgical c-section

SECONDARY OUTCOMES:
dosage of vasopressors administered | day one
  vasopressors administered during surgery
number of episodes of nausea | 24 hours after surgery
occurrence & intensity of itching | 24 hours after surgery
pain scores reported by the patient | 24 hours after surgery
dosage of anticholinergics administered | 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Hackworth, MD, Principal Investigator — University of Virginia Anesthesiology
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Hawkins JL. Anesthesia-related maternal mortality. Clin Obstet Gynecol. 2003 Sep;46(3):679-87. doi: 10.1097/00003081-200309000-00020. No abstract available. PMID 12972749
- [Background] Mhyre JM, Riesner MN, Polley LS, Naughton NN. A series of anesthesia-related maternal deaths in Michigan, 1985-2003. Anesthesiology. 2007 Jun;106(6):1096-104. doi: 10.1097/01.anes.0000267592.34626.6b. PMID 17525583
- [Background] Lee LA, Posner KL, Domino KB, Caplan RA, Cheney FW. Injuries associated with regional anesthesia in the 1980s and 1990s: a closed claims analysis. Anesthesiology. 2004 Jul;101(1):143-52. doi: 10.1097/00000542-200407000-00023. PMID 15220784
- [Background] Liu SS, McDonald SB. Current issues in spinal anesthesia. Anesthesiology. 2001 May;94(5):888-906. doi: 10.1097/00000542-200105000-00030. No abstract available. PMID 11388543
- [Background] Jackson R, Reid JA, Thorburn J. Volume preloading is not essential to prevent spinal-induced hypotension at caesarean section. Br J Anaesth. 1995 Sep;75(3):262-5. doi: 10.1093/bja/75.3.262. PMID 7547039
- [Background] Kinsella SM, Lohmann G. Supine hypotensive syndrome. Obstet Gynecol. 1994 May;83(5 Pt 1):774-88. PMID 8164943
- [Background] Rout CC, Rocke DA. Prevention of hypotension following spinal anesthesia for cesarean section. Int Anesthesiol Clin. 1994 Spring;32(2):117-35. No abstract available. PMID 8063445
- [Background] Mathru M, Rao TL, Kartha RK, Shanmugham M, Jacobs HK. Intravenous albumin administration for prevention of spinal hypotension during cesarean section. Anesth Analg. 1980 Sep;59(9):655-8. PMID 7191222
- [Background] Dahlgren G, Granath F, Pregner K, Rosblad PG, Wessel H, Irestedt L. Colloid vs. crystalloid preloading to prevent maternal hypotension during spinal anesthesia for elective cesarean section. Acta Anaesthesiol Scand. 2005 Sep;49(8):1200-6. doi: 10.1111/j.1399-6576.2005.00730.x. PMID 16095463
- [Background] Ueyama H, He YL, Tanigami H, Mashimo T, Yoshiya I. Effects of crystalloid and colloid preload on blood volume in the parturient undergoing spinal anesthesia for elective Cesarean section. Anesthesiology. 1999 Dec;91(6):1571-6. doi: 10.1097/00000542-199912000-00006. PMID 10598596
- [Background] Riley ET, Cohen SE, Rubenstein AJ, Flanagan B. Prevention of hypotension after spinal anesthesia for cesarean section: six percent hetastarch versus lactated Ringer's solution. Anesth Analg. 1995 Oct;81(4):838-42. doi: 10.1097/00000539-199510000-00031. PMID 7574020
- [Background] Campagna JA, Carter C. Clinical relevance of the Bezold-Jarisch reflex. Anesthesiology. 2003 May;98(5):1250-60. doi: 10.1097/00000542-200305000-00030. No abstract available. PMID 12717149
- [Background] Villalon CM, Centurion D. Cardiovascular responses produced by 5-hydroxytriptamine:a pharmacological update on the receptors/mechanisms involved and therapeutic implications. Naunyn Schmiedebergs Arch Pharmacol. 2007 Oct;376(1-2):45-63. doi: 10.1007/s00210-007-0179-1. Epub 2007 Aug 17. PMID 17703282
- [Background] Veelken R, Sawin LL, DiBona GF. Epicardial serotonin receptors in circulatory control in conscious Sprague-Dawley rats. Am J Physiol. 1990 Feb;258(2 Pt 2):H466-72. doi: 10.1152/ajpheart.1990.258.2.H466. PMID 2309912
- [Background] Owczuk R, Wenski W, Polak-Krzeminska A, Twardowski P, Arszulowicz R, Dylczyk-Sommer A, Wujtewicz MA, Sawicka W, Morzuch E, Smietanski M, Wujtewicz M. Ondansetron given intravenously attenuates arterial blood pressure drop due to spinal anesthesia: a double-blind, placebo-controlled study. Reg Anesth Pain Med. 2008 Jul-Aug;33(4):332-9. doi: 10.1016/j.rapm.2008.01.010. PMID 18675744
- [Background] Martinek RM. Witnessed asystole during spinal anesthesia treated with atropine and ondansetron: a case report. Can J Anaesth. 2004 Mar;51(3):226-30. doi: 10.1007/BF03019100. PMID 15010403
- [Background] FDA Prescribing Information. Web retrieved 7/8/2009 .http://www.fda.org
- [Background] Tucker ML, Jackson MR, Scales MD, Spurling NW, Tweats DJ, Capel-Edwards K. Ondansetron: pre-clinical safety evaluation. Eur J Cancer Clin Oncol. 1989;25 Suppl 1:S79-93. PMID 2533905
- [Background] Einarson A, Maltepe C, Navioz Y, Kennedy D, Tan MP, Koren G. The safety of ondansetron for nausea and vomiting of pregnancy: a prospective comparative study. BJOG. 2004 Sep;111(9):940-3. doi: 10.1111/j.1471-0528.2004.00236.x. PMID 15327608
- [Background] Sullivan CA, Johnson CA, Roach H, Martin RW, Stewart DK, Morrison JC. A pilot study of intravenous ondansetron for hyperemesis gravidarum. Am J Obstet Gynecol. 1996 May;174(5):1565-8. doi: 10.1016/s0002-9378(96)70607-5. PMID 9065130
- [Background] Kuscu NK, Koyuncu F. Hyperemesis gravidarum: current concepts and management. Postgrad Med J. 2002 Feb;78(916):76-9. doi: 10.1136/pmj.78.916.76. PMID 11807187
- [Background] Asker C, Norstedt Wikner B, Kallen B. Use of antiemetic drugs during pregnancy in Sweden. Eur J Clin Pharmacol. 2005 Dec;61(12):899-906. doi: 10.1007/s00228-005-0055-1. Epub 2005 Nov 18. PMID 16328314
- [Background] Phillips TW Jr, Broussard DM, Sumrall WD 3rd, Hart SR. Intraoperative oxygen administration does not reduce the incidence or severity of nausea or vomiting associated with neuraxial anesthesia for cesarean delivery. Anesth Analg. 2007 Oct;105(4):1113-7, table of contents. doi: 10.1213/01.ane.0000278626.54116.0e. PMID 17898396
- [Background] Siddik-Sayyid SM, Aouad MT, Taha SK, Azar MS, Hakki MA, Kaddoum RN, Nasr VG, Yazbek VG, Baraka AS. Does ondansetron or granisetron prevent subarachnoid morphine-induced pruritus after cesarean delivery? Anesth Analg. 2007 Feb;104(2):421-4. doi: 10.1213/01.ane.0000253668.10453.de. PMID 17242102
- [Background] Yeh HM, Chen LK, Lin CJ, Chan WH, Chen YP, Lin CS, Sun WZ, Wang MJ, Tsai SK. Prophylactic intravenous ondansetron reduces the incidence of intrathecal morphine-induced pruritus in patients undergoing cesarean delivery. Anesth Analg. 2000 Jul;91(1):172-5. doi: 10.1097/00000539-200007000-00032. PMID 10866907
- [Background] Yazigi A, Chalhoub V, Madi-Jebara S, Haddad F, Hayek G. Prophylactic ondansetron is effective in the treatment of nausea and vomiting but not on pruritus after cesarean delivery with intrathecal sufentanil-morphine. J Clin Anesth. 2002 May;14(3):183-6. doi: 10.1016/s0952-8180(01)00381-6. PMID 12031749
- [Background] Sarvela PJ, Halonen PM, Soikkeli AI, Kainu JP, Korttila KT. Ondansetron and tropisetron do not prevent intraspinal morphine- and fentanyl-induced pruritus in elective cesarean delivery. Acta Anaesthesiol Scand. 2006 Feb;50(2):239-44. doi: 10.1111/j.1399-6576.2006.00934.x. PMID 16430549
- [Background] Abouleish EI, Rashid S, Haque S, Giezentanner A, Joynton P, Chuang AZ. Ondansetron versus placebo for the control of nausea and vomiting during Caesarean section under spinal anaesthesia. Anaesthesia. 1999 May;54(5):479-82. doi: 10.1046/j.1365-2044.1999.00798.x. PMID 10995148
- [Background] George RB, Allen TK, Habib AS. Serotonin receptor antagonists for the prevention and treatment of pruritus, nausea, and vomiting in women undergoing cesarean delivery with intrathecal morphine: a systematic review and meta-analysis. Anesth Analg. 2009 Jul;109(1):174-82. doi: 10.1213/ane.0b013e3181a45a6b. PMID 19535708
- [Background] Tang J, Wang B, White PF, Watcha MF, Qi J, Wender RH. The effect of timing of ondansetron administration on its efficacy, cost-effectiveness, and cost-benefit as a prophylactic antiemetic in the ambulatory setting. Anesth Analg. 1998 Feb;86(2):274-82. doi: 10.1097/00000539-199802000-00010. PMID 9459232
- [Derived] Terkawi AS, Tiouririne M, Mehta SH, Hackworth JM, Tsang S, Durieux ME. Ondansetron Does Not Attenuate Hemodynamic Changes in Patients Undergoing Elective Cesarean Delivery Using Subarachnoid Anesthesia: A Double-Blind, Placebo-Controlled, Randomized Trial. Reg Anesth Pain Med. 2015 Jul-Aug;40(4):344-8. doi: 10.1097/AAP.0000000000000274. PMID 26066384